CLINICAL TRIAL: NCT01177683
Title: A Phase I/II Trial of Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin in Patients With Relapsed or Refractory Multiple Myeloma: Hoosier Cancer Research Network MM08-141
Brief Title: Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin for Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Sherif Farag, MB, BS (Other)
Collaborators: Hoosier Cancer Research Network (Other); Cephalon, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sherif Farag, MB, BS, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM08-141
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Doxorubicin; Bortezomib; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Bendamustine in combination with bortezomib and pegylated liposomal doxorubicin.
  Interventions: Drug: Bendamustine; Drug: Doxorubicin; Drug: Bortezomib; Drug: Filgrastim

INTERVENTIONS:
Drug: Bendamustine — Phase I component:
  Bendamustine escalating cohorts to determine MTD, IV over 1 hour, Days 1 and 4
Drug: Doxorubicin — Phase I and II components:
  Pegylated liposomal doxorubicin, 30 mg/m2 IV over 1 hour, Day 4
Drug: Bortezomib — Phase I and II components:
  Bortezomib 1.3 mg/m2 IV bolus, Days 1, 4, 8, and 11
Drug: Bendamustine — Phase II component:
  Bendamustine at at MTD IV over 1 hour, Days 1 and 4
Drug: Filgrastim — Phase II component:
  Filgrastim (if defined in MTD) 5 µg/kg/day SC, starting day 6 until neutrophil recovery to ANC >1000

SUMMARY:
This is an open label phase I/II trial to determine the safety and the biologic activity of the bendamustine, bortezomib and pegylated liposomal doxorubicin combination.

DETAILED DESCRIPTION:
Phase I component Bortezomib 1.3 mg/m2 IV bolus, Days 1, 4, 8, and 11 Doxorubicin 30 mg/m2 IV over 1 hour, Day 4 Bendamustine escalating cohorts IV over 1 hour, Days 1 and 4 1 Cycle = 28 days

Phase II component Bortezomib 1.3 mg/m2 IV bolus, Days 1, 4, 8, and 11 Doxorubicin 30 mg/m2 IV over 1 hour, Day 4 Bendamustine at MTD IV over 1 hour, Days 1 and 4 Filgrastim (if defined in MTD) 5 µg/kg/day SC, Starting day 6 until neutrophil recovery to ANC >1000

1 Cycle = 28 days; Patients will continue treatment for a total of up to 8 cycles.

ECOG Performance Status: 0-2

Hematopoietic:

* Absolute neutrophil count (ANC) ≥ 1.2 x K/mm3
* Platelets ≥ 75 x K/mm3

Hepatic:

* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* AST ≤ 2.5 x ULN
* ALT ≤ 2.5 x ULN

Renal:

* Serum creatinine < 3.0 mg/dL

Cardiovascular:

* LVEF >45% corrected by MUGA scan or echocardiogram.
* No unstable angina pectoris or recent myocardial infarction (within 6 months)

ELIGIBILITY:
Inclusion Criteria:

* A histologically established diagnosis of multiple myeloma with evidence of relapse or refractory disease.
* Must have a detectable serum or urine M-Protein by protein electrophoresis that is at least 500 mg/dL (serum) or 1 gm/24 hours (urine), respectively, or serum free light chain level >100 mg/l for the involved free light chain.
* Must have received at least one (1) prior line of systemic treatment that has included either lenalidomide or thalidomide.
* Must be willing to provide correlative blood samples.

Exclusion Criteria:

* Must not have received an excessive cumulative dose of anthracycline
* No ≥ grade 2 peripheral neuropathy.
* No cytotoxic chemotherapy within 30 days prior to registration for protocol therapy.
* No autologous stem cell transplant within 6 months prior to registration for protocol therapy
* No prior radiation therapy to > 25% of bone marrow forming bones (i.e., pelvis) within 30 days prior to registration for protocol therapy. See Study Procedures Manual to calculate percent of prior radiation.
* No current corticosteroid therapy in doses greater than 10 mg daily of prednisone (or equivalent) if given for management of co-morbid conditions.
* No known central nervous system involvement by myeloma.
* No poorly controlled intercurrent illness including, but not limited to, ongoing or active infection, poorly controlled diabetes, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social climate that in the opinion of the investigator would limit compliance with study requirements.
* No patients known to be positive for HIV, or active Hepatitis A, B, or C.
* No major surgery within 30 days prior to registration for protocol therapy. Placement of a venous access device within 30 days prior to registration for protocol therapy is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, M.B., B.S., Study Chair — Hoosier Cancer Research Network
Locations (7):
- United States (7):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - IU Health Arnett Cancer Center, Lafayette, Indiana
  - Metro Health Cancer Care, Wyoming, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio

REFERENCES:
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Level 1 : Bendamustine at 90mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin.: Bendamustine: At Phase I level I, Bendamustine will be administered at 90 mg/m^2 by IV over 1 hour at days 1 and 4 of the 28 day treatment cycle.
  Filgrastim (if defined in MTD) will be administered at 5 µg/kg/day SC, starting day 6 until neutrophil recovery to ANC >1000.
  Doxorubicin:
  Pegylated liposomal doxorubicin at phase I will be administered at 30 mg/m2 by IV over 1 hour, at day 4 of the 28 day treatment cycle.
  Bortezomib:
  Bortezomib at Phase I will be administered at 1.3 mg/m2 by IV bolus on days 1, 4, 8, and 11 of the 28 day cycle.
- Phase I Level 2 : Bendamustine at 120mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin.: Bendamustine: At Phase I level 2, Bendamustine will be administered at 120 mg/m^2 by IV over 1 hour at days 1 and 4 of the 28 day treatment cycle.
  Filgrastim (if defined in MTD) will be administered at 5 µg/kg/day SC, starting day 6 until neutrophil recovery to ANC >1000.
  Doxorubicin:
  Pegylated liposomal doxorubicin at phase I will be administered at 30 mg/m2 by IV over 1 hour, at day 4 of the 28 day treatment cycle.
  Bortezomib:
  Bortezomib at Phase I will be administered at 1.3 mg/m2 by IV bolus on days 1, 4, 8, and 11 of the 28 day cycle.
- Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.: Bendamustine:
  At phase II, Bendamustine will be administered at 90mg/m^2 by IV over 1 hour at days 1 and 4 of the 28 day treatment cycle.
  Doxorubicin:
  Pegylated liposomal doxorubicin at phase II will be administered at 30 mg/m2 by IV over 1 hour, at day 4 of the 28 day treatment cycle.
  Bortezomib:
  Bortezomib at Phase II will be administered at 1.3 mg/m2 by IV bolus or SQ injection on days 1, 4, 8, and 11 of the 28 day cycle.
Period: Study Treatment
Arm/Group | Phase I Level 1 : Bendamustine at 90mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase I Level 2 : Bendamustine at 120mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.
Started | 3 | 3 | 26
Completed | 0 | 0 | 2
Not Completed | 3 | 3 | 24
Not completed — Disease Progressions during treatment | 2 | 0 | 3
Not completed — Adverse Event | 0 | 1 | 12
Not completed — Patient Withdrawal After Therapy Start | 0 | 2 | 1
Not completed — Alternative therapy | 0 | 0 | 4
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Patient withdrawal before therapy start | 0 | 0 | 1
Not completed — Symptomatic Deterioration | 0 | 0 | 1
Not completed — Subject came off study without receiving any treatment. | 0 | 0 | 1
Period: Follow up
Arm/Group | Phase I Level 1 : Bendamustine at 90mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase I Level 2 : Bendamustine at 120mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.
Started | 3 | 3 | 24
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 24
Not completed — Patient lost to follow up | 0 | 0 | 2
Not completed — Death | 2 | 1 | 7
Not completed — Study closed by Sponsor due slow enrollment. | 1 | 2 | 15

BASELINE CHARACTERISTICS:
Groups:
- Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.: Bendamustine:
  At phase II, Bendamustine will be administered at 90mg/m^2 by IV over 1 hour at days 1 and 4 of the 28 day treatment cycle.
  Doxorubicin:
  Pegylated liposomal doxorubicin at phase II will be administered at 30 mg/m2 by IV over 1 hour,at day 4 of the 28 day treatment cycle.
  Bortezomib:
  Bortezomib at Phase II will be administered at 1.3 mg/m2 by IV bolus or SQ injection on days 1, 4, 8, and 11 of the 28 day cycle.
- Total: Total of all reporting groups
Arm/Group | Phase I Level 1 : Bendamustine at 90mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase I Level 2 : Bendamustine at 120mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin. | Total
Number analyzed (Participants) | 3 | 3 | 26 | 32
Age, Continuous [Mean (Full Range); unit: years] | 61.67 [52 to 70] | 53.33 [41 to 69] | 62.58 [44 to 89] | 61.63 [41 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 11 | 15
  Male | 1 | 1 | 15 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 25 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 4
  White | 3 | 1 | 23 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
ECOG Performance Status (Baseline [Count of Participants; unit: Participants] — ECOG PERFORMANCE STATUS:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 1 | 2 | 13 | 16
    1 | 2 | 1 | 11 | 14
    2 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase I: MTD of Bendamustine When Combined With Bortezomib and Pegylated Liposomal Doxorubicin.
Description: In the first phase, MTD of bendamustine was determined in combination with bortezomib and pegylated liposomal doxorubicin to gain a better idea of safe dosing before proceeding with the second phase to assess efficacy. Assuming myelosuppression being a dose-limiting effect that could have been overcome with growth factor support, MTD of the combination with myeloid growth factor support was also tested.
Time Frame: From C1D1 up to a maximum of 7 months or until death
Measure: Number; unit: mg/m^2
Groups:
- Phase I Level 1:Bendamustine at 90 mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin.: Bendamustine: At Phase I level 1, Bendamustine will be administered at 90 mg/m^2 by IV over 1 hour at days 1 and 4 of the 28 day treatment cycle.
  Filgrastim (if defined in MTD) will be administered at 5 µg/kg/day SC, starting day 6 until neutrophil recovery to ANC >1000.
  Doxorubicin:
  Pegylated liposomal doxorubicin at phase I will be administered at 30 mg/m2 by IV over 1 hour, at day 4 of the 28 day treatment cycle.
  Bortezomib:
  Bortezomib at Phase I will be administered at 1.3 mg/m2 by IV bolus on days 1, 4, 8, and 11 of the 28 day cycle.
- Phase I Level 2:Bendamustine at 120 mg/m^2 With Bortezomib and Pegylated Liposomal: Bendamustine: At Phase I level 2, Bendamustine will be administered at 120 mg/m^2 by IV over 1 hour at days 1 and 4 of the 28 day treatment cycle.
  Filgrastim (if defined in MTD) will be administered at 5 µg/kg/day SC, starting day 6 until neutrophil recovery to ANC >1000.
  Doxorubicin:
  Pegylated liposomal doxorubicin at phase I will be administered at 30 mg/m2 by IV over 1 hour, at day 4 of the 28 day treatment cycle.
  Bortezomib:
  Bortezomib at Phase I will be administered at 1.3 mg/m2 by IV bolus on days 1, 4, 8, and 11 of the 28 day cycle.
Arm/Group | Phase I Level 1:Bendamustine at 90 mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase I Level 2:Bendamustine at 120 mg/m^2 With Bortezomib and Pegylated Liposomal
Number analyzed (Participants) | 3 | 3
mg/m^2 | 120 | 120

2. Primary Outcome: Phase II : Overall Response Rate
Description: Overall response rate (CR+PR) of bendamustine in association with bortezomib and pegylated liposomal doxorubicin was assessed in patients with relapsed or refractory Multiple Myeloma. Per modified International Myeloma Working Group criteria: Complete Response (CR) : Negative for monoclonal protein by immunofixation on the serum and urine, and Disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow ; PR : 50% or more reduction in serum M-protein and 90% or more reduction in urine M-protein or to <200 mg/24hours or a 50% or more reduction in free light chain level ; Overall Response (OR) = CR +PR.
Time Frame: From C1D1 up to a maximum of 52 months or until death
Population: Two subjects never received treatment. Therefore, they were not included in any assessment of objectives.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.
Number analyzed (Participants) | 24
Participants
  CR+PR | 14
  Non-CR+PR | 9
  Missing | 1

3. Secondary Outcome: Phase I & Phase II : Toxicity of Treatment Regimen
Description: Toxicity profile (for all patients) were presented by rate of overall toxicity and rates of grade 3 or 4 toxicities analyzed separately and combined.
Time Frame: From C1D1 until death or up to a maximum of 54 months
Population: Two subjects in phase II never received treatment. Therefore, they were not included in any assessment of objectives.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Level 1 : Bendamustine at 90mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase I Level 2 : Bendamustine at 120mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.
Number analyzed (Participants) | 3 | 3 | 24
Participants
  Number of patients had at least one adverse event of any grade | 3 | 3 | 24
  Number of patients had at least one grade 3 or greater adverse event | 2 | 3 | 19
  Number of patients had at least one grade 3 or greater treatment related adverse event | 2 | 3 | 14
  Number of patients having serious adverse event | 1 | 1 | 8

4. Secondary Outcome: Phase II : Time to Progression
Description: The time from the start of treatment (i.e., first dose) of MM patients treated with bendamustine, bortezomib and pegylated liposomal doxorubicin to disease progression, with disease progression and death due to disease progression as events and deaths due to causes other than progression as censored. Censoring date will be the last disease evaluation date for patient without progression/death or date of death due to other diseases for patients' deaths due to other causes.Per modified International Myeloma Working Group criteria: Progressive disease (PD) is reported if any one of the following criteria is met:
  Increase of 25% or more in serum or urine M-protein from baseline;Serum M-protein and/or the absolute increase must be ≥0.5 g/dL;Urine M-protein and/or absolute increase must be ≥200 mg/24 hours ; Development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas;Development of hyperc.
Time Frame: From C1D1 up to a maximum of 54 months or until death
Population: Two subjects never received treatment. Therefore, they were not included in any assessment of objectives.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.
Number analyzed (Participants) | 24
months | 20.53 [6.47 to 27.47]

5. Secondary Outcome: Phase II: Progression-free Survival (PFS)
Description: The time from the start of treatment of MM patients treated with bendamustine, bortezomib and pegylated liposomal doxorubicin. to disease progression or death (regardless of cause of death), whichever comes first. Censoring date will be the last disease evaluation date.Per modified International Myeloma Working Group criteria: Progressive disease (PD) is reported if any one of the following criteria is met:
  Increase of 25% or more in serum or urine M-protein from baseline;Serum M-protein and/or the absolute increase must be ≥0.5 g/dL;Urine M-protein and/or absolute increase must be ≥200 mg/24 hours ; Development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas;Development of hyperc.
Time Frame: From C1D1 up to a maximum of 54 months until death
Population: Two subjects never received treatment. Therefore, they were not included in any assessment of objectives.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.
Number analyzed (Participants) | 24
months | 18.96 [6.47 to 26.91]

6. Secondary Outcome: Phase II: Duration of Survival
Description: Duration of MM patients treated with bendamustine, bortezomib and pegylated liposomal doxorubicin. from first date of at least partial response to the time of progression or death due to disease progression as events, with disease progression and death due to disease progression as events and deaths due to causes other than progression as censored. Censoring date will be the last disease evaluation date or date of death due to other causes as appropriate.
Time Frame: From C1D1 up to a maximum of 52 months
Population: Two subjects never received treatment. Therefore, they were not included in any assessment of objectives.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.
Number analyzed (Participants) | 24
months | 13.80 [7.85 to NA] — The upper limit could not be determined within 95% confidence interval due to low enrollment.The limited sample size is not enough to accurately estimate the upper limit of the confidence interval. A larger sample size would be needed to get a more reliable estimate.

7. Secondary Outcome: Phase II: Overall Survival
Description: The time from the start of treatment to death from any cause with last date known alive as censoring date.
Time Frame: From C1D1 up to a maximum of 54 months or until death
Population: Two subjects never received treatment. Therefore, they were not included in any assessment of objectives.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.
Number analyzed (Participants) | 24
months | 30.13 [9.69 to NA] — The upper limit could not be determined within 95% confidence interval due to low enrollment.The limited sample size is not enough to accurately estimate the upper limit of the confidence interval. A larger sample size would be needed to get a more reliable estimate.

ADVERSE EVENTS:
Time Frame: From C1D1 up to at least 30 days after final protocol treatment or up to a maximum of 54 months.
Description: Adverse events will be recorded from the time of consent and for at least 30 days after final protocol treatment.
  SAEs must be reported during the course of the study within 24 hours of discovery of the event.
Arm/Group | Phase I Level 1 : Bendamustine at 90mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase I Level 2 : Bendamustine at 120mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin.
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3 | 7/26
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 8/26
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Level 1 : Bendamustine at 90mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. (N=3) | Phase I Level 2 : Bendamustine at 120mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. (N=3) | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin. (N=26)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Colon (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
ENTERITIS (INFLAMMATION OF THE SMALL BOWEL) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
HYPOTENSION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
INFECTION (MENINGITIS) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - LUNG (PNEUMONIA) (Infections and infestations) | 0 (0) | 0 (0) | 2 (4)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - UPPER AIRWAY NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Level 1 : Bendamustine at 90mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. (N=3) | Phase I Level 2 : Bendamustine at 120mg/m^2 With Bortezomib and Pegylated Liposomal Doxorubicin. (N=3) | Phase II : Bendamustine in Combination With Bortezomib and Pegylated Liposomal Doxorubicin. (N=26)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Anorexia (Gastrointestinal disorders) | 2 (3) | 3 (4) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 3 (3) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (4) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (5) | 3 (6) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1) | 1 (4) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (17) | 1 (5) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (19) | 2 (8) | 0 (0)
Mucositis/stomatitis (clinical exam) - Esophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-upper (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 3 (4) | 0 (0)
Neuropathy: sensory (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (11) | 1 (2) | 0 (0)
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0)
Pain - Back (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Pain - Bone (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pain - Extremity-limb (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Pain - Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Head/headache (Nervous system disorders) | 2 (6) | 0 (0) | 0 (0)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Oral cavity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 1 (7) | 2 (4) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (4) | 1 (2) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 1 (1) | 2 (4) | 0 (0)
Trismus (difficulty, restriction or pain when opening mouth) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (5) | 0 (0)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Weight loss (General disorders) | 1 (2) | 0 (0) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Infection - Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Pain - Other (Specify, __) (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Sweating (diaphoresis) (General disorders) | 0 (0) | 1 (2) | 0 (0)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (9)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 0 (0) | 0 (0) | 5 (5)
ALLERGY/IMMUNOLOGY - OTHER (SPECIFY, __) (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4)
ANOREXIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (12)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (6)
AUDITORY/EAR - OTHER (SPECIFY, __) (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
BILIRUBIN (HYPERBILIRUBINEMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
BRUISING (IN ABSENCE OF GRADE 3 OR 4 THROMBOCYTOPENIA) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTEREMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
CONFUSION (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (8)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 6 (9)
CREATININE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (10)
DEHYDRATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 13 (32)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
DRY EYE SYNDROME (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5)
EDEMA:HEAD AND NECK (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
EDEMA:LIMB (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4)
ENDOCRINE - OTHER (SPECIFY, __) (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 0 (0) | 0 (0) | 18 (42)
FEBRILE NEUTROPENIA (Infections and infestations) | 0 (0) | 0 (0) | 5 (7)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 0 (0) | 0 (0) | 3 (6)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
GLOMERULAR FILTRATION RATE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (8)
HEMOGLOBIN (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 10 (36)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (6)
HEMORRHAGE, GI - ANUS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
HEMORRHAGE/BLEEDING - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4)
HYPOTENSION (Cardiac disorders) | 0 (0) | 0 (0) | 2 (4)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
INFECTION- SKIN (CELLULITIS) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - DUODENUM (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - MUCOSA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - NERVE-PERIPHERAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - ORAL CAVITY-GUMS (GINGIVITIS) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SINUS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SKIN (CELLULITIS) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - UPPER AERODIGESTIVE NOS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - UPPER AIRWAY NOS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - URINARY TRACT NOS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
INFECTION WITH UNKNOWN ANC - SKIN (CELLULITIS) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE REACTION/EXTRAVASATION CHANGES (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6)
INR (INTERNATIONAL NORMALIZED RATIO OF PROTHROMBIN TIME) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
INSOMNIA (General disorders) | 0 (0) | 0 (0) | 5 (6)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (31)
LYMPHATICS - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (23)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
METABOLIC/LABORATORY - OTHER (SPECIFY, __) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
MOOD ALTERATION - AGITATION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
MOOD ALTERATION - ANXIETY (Nervous system disorders) | 0 (0) | 0 (0) | 4 (5)
MOOD ALTERATION - DEPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ESOPHAGUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ORAL CAVITY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (5)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - ESOPHAGUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - ORAL CAVITY (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 20 (30)
NEUROLOGY - OTHER (SPECIFY, __) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (4)
NEUROPATHY: SENSORY (Nervous system disorders) | 0 (0) | 0 (0) | 14 (23)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 12 (41)
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
PAIN - BACK (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (4)
PAIN - BONE (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (5)
PAIN - CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN - EXTREMITY-LIMB (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 6 (7)
PAIN - HEAD/HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 4 (5)
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (6)
PAIN - MUSCLE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN - NECK (General disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN - OTHER (SPECIFY, __) (General disorders) | 0 (0) | 0 (0) | 3 (5)
PAIN - PAIN NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN - THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PHLEBITIS (INCLUDING SUPERFICIAL THROMBOSIS) (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
PLATELETS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 13 (40)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (11)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (8)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (11)
SOMNOLENCE/DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - ATRIAL TACHYCARDIA/PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (FAINTING) (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ULCER, GI - ESOPHAGUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
VASCULAR - OTHER (SPECIFY, __) (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
VISION-BLURRED VISION (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (14)
WEIGHT LOSS (General disorders) | 0 (0) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT01177683/Prot_SAP_000.pdf